CLINICAL TRIAL: NCT04730154
Title: The Effect of Perceived Injustice Targeted Pain Neuroscience Education and Motivational Interviewing Compared to Biomedical Focused Education in Breast Cancer Survivors
Brief Title: PI-targeted PNE+MI Compared to BIOMEDICAL Education in BCS
Acronym: BCS-PI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); Kom Op Tegen Kanker (Other); Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANI251_BCS-PI
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Survivorship; Pain, Chronic
Keywords: Breast cancer survivor; Perceived injustice; Pain Neuroscience Education; Motivational Interviewing; Biomedical Education
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Neuroscience Education (PNE) + Motivational Interviewing (MI) (Experimental): Breast cancer survivors assigned to the experimental intervention will participate in 1 online PNE session followed by 3 PNE + MI sessions spread over 4 weeks. Each session will last for approximately 45 minutes and all sessions will be held in one-on-one format, allowing to individually tailor content to the patient's maladaptive beliefs and perceived injustice. After the first live session, breast cancer survivors will receive a perceived injustice-targeted PNE information leaflet that they need to read carefully at home.
  Interventions: Behavioral: Pain Neuroscience Education (PNE); Behavioral: Motivational Interviewing (MI)
- Biomedically-focused Education (Active Comparator): Breast cancer survivors assigned to the experimental intervention will participate in 1 online biomedically-focused education session followed by 3 biomedically-focused education sessions spread over 4 weeks. Each session will last for approximately 45 minutes and all sessions will be held in one-on-one format in order to balance nonspecific treatment effects between treatment arms, the duration, format and number of sessions as well as the didactical approach will be identical in both treatment groups. After the first live session, breast cancer survivors will receive an information leaflet from 'Kom op tegen Kanker' regarding 'Pain in and after treatment' that they need to read carefully at home.
  Interventions: Behavioral: Biomedically-focused education

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE) — PNE is a cognitive behavioural intervention, including educating patients that pain is an output product of the brain resulting from input from multiple central and peripheral nervous system processes and leading to threat perception. Transferring that knowledge to patients, allows them to understand, accept and effectively cope with their pain. In order to obtain the targeted behavioural change, motivational interviewing is used as the communication process throughout PNE.
  Arms: Pain Neuroscience Education (PNE) + Motivational Interviewing (MI)
Behavioral: Motivational Interviewing (MI) — Motivational interviewing is a directive, collaborative, patient-centered communication approach for eliciting and enhancing motivation for behaviour change by helping clients to resolve ambivalence and uncertainty.
  Arms: Pain Neuroscience Education (PNE) + Motivational Interviewing (MI)
Behavioral: Biomedically-focused education — The traditional biomedical-focused education programme explains patient's pain experience from a tissue (injured versus healthy tissue) and biomechanical perspective.
  Arms: Biomedically-focused Education

SUMMARY:
Breast cancer is the most frequently diagnosed cancer in women worldwide. An important portion of the breast cancer survivors will face chronic pain complaints. These pain complaints do not only impact the patient's quality of life but also prevents resumption of activities, leading to huge economic costs. 30% of all breast cancer survivors with pain present with perceived injustice which has been conceptualized as a multidimensional appraisal process characterized by a tendency to interpret one's losses as severe and irreparable, to attribute blame to others for one's suffering and to experience a sense of unfairness. Perceived injustice is also associated with increased opioid prescription and use, urging the need for targeted interventions to diminish perceived injustice.

Despite the fact that specific treatment plans for perceived injustice are not yet proven, pain neuroscience education (PNE) is proven to reassure and encourage towards activity. In order to obtain the targeted behavioural change, motivational interviewing (MI) is used as the communication process throughout PNE.

A multi-centre, parallel, two-arm, investigator-blinded study with 4-weeks intervention and two years follow-up will be conducted in 156 BCS with PI and pain. These will be randomly assigned to the intervention or usual care group. The groups will receive 1 online session, an information leaflet and 3 live sessions of education spread over 4 weeks. Pain neuroscience education in combination with motivational interviewing will be given in the experimental group and biomedically-focused education to the control group.

The primary scientific objective of the study is to examine whether perceived injustice-targeted PNE is superior to biomedically-focused pain education in reducing pain after 12 months in breast cancer survivors with perceived injustice and pain.

The secondary objectives of the study are to examine whether perceived injustice-targeted PNE, compared to biomedically-focused pain education, results in improving health-related quality of life, reducing perceived injustice and opioid use after 24 months in breast cancer survivors with perceived injustice and pain, and to conduct a health-care cost analysis which will finally result in a recommendation concerning the use of perceived injustice-targeted PNE in breast cancer survivors with perceived injustice and pain.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible, participants have to fulfil the definition for survivorship introduced by the European Organisation of Research and Treatment of Cancer (EORTC) Survivorship Task Force, in which a cancer survivor is: 'any person who has been diagnosed with cancer, has completed his or her primary treatment (with the exception of maintenance therapy) and has no evidence of active disease'. Therefore, participants need to:

1. Be women aged 18 years or older.
2. Be in complete remission and should have finished their primary treatment with a curative intent at least 3 months prior to study participation. Adjuvant hormonal therapy and immunotherapy are tolerated.
3. Report a pain severity of at least 3/10 on the Brief Pain Inventory.
4. Be able to speak and read Dutch in order to give informed consent and to complete the assessment tools.
5. Show evidence of perceived injustice, defined as a score of 17 or higher on the Injustice Experience Questionnaire (IEQ).

Exclusion Criteria

Participants will be excluded if they:

1. Are diagnosed with new neoplasms or metastases.
2. Have not reached the stable level of a chronic disease and/or which is causing pain complaints (e.g. fibromyalgia, rheumatoid arthritis…).
3. Are suffering from severe psychological or psychiatric diseases.
4. Are suffering from dementia or cognitive impairment (unable to understand the test instructions and/or a result of ≤11, corresponding with MMSE ≤23, on the Six-item Cognitive Impairment Test (6-item CIT) is a short questionnaire containing 6 items.
5. Recently started a new therapy which has not yet resulted in a stable level and might interference with one of the treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 156 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain Outcome | T0: within the week before the randomisation and the start of the intervention
  The Brief Pain Inventory is a 14-item questionnaire assessing worst pain, pain severity, and pain interference in cancer patients over the past week, reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The Brief Pain Inventory is the most common, reliable and valid outcome measure to assess pain in cancer survivors (Cronbach's alfa and test-retest reliability score > 0.80).
Pain Outcome | T1: immediately after completing intervention
  The Brief Pain Inventory is a 14-item questionnaire assessing worst pain, pain severity, and pain interference in cancer patients over the past week, reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The Brief Pain Inventory is the most common, reliable and valid outcome measure to assess pain in cancer survivors (Cronbach's alfa and test-retest reliability score > 0.80).
Pain Outcome | T2: 6 months after therapy completion
  The Brief Pain Inventory is a 14-item questionnaire assessing worst pain, pain severity, and pain interference in cancer patients over the past week, reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The Brief Pain Inventory is the most common, reliable and valid outcome measure to assess pain in cancer survivors (Cronbach's alfa and test-retest reliability score > 0.80).
Pain Outcome | T3: 12 months after therapy completion
  The Brief Pain Inventory is a 14-item questionnaire assessing worst pain, pain severity, and pain interference in cancer patients over the past week, reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The Brief Pain Inventory is the most common, reliable and valid outcome measure to assess pain in cancer survivors (Cronbach's alfa and test-retest reliability score > 0.80).
Pain Outcome | T4: 24 months after therapy completion
  The Brief Pain Inventory is a 14-item questionnaire assessing worst pain, pain severity, and pain interference in cancer patients over the past week, reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The Brief Pain Inventory is the most common, reliable and valid outcome measure to assess pain in cancer survivors (Cronbach's alfa and test-retest reliability score > 0.80).

SECONDARY OUTCOMES:
Health-related quality of life (HR-QoL) | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) is a 30-item cancer-specific questionnaire developed for the assessment of quality of life in cancer patients. The EORTC QLQ-C30 is widely used in cancer studies, has been translated and validated in over 100 languages and shows acceptable psychometric properties. The internal consistence measured by Cronbach's resulted in 0.94.
Perceived injustice (PI) | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  The 12-item Injustice Experience Questionnaire (IEQ) will be used to assess perceived injustice. Participants have to rate the frequency of 12 different pain-related statements on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time). The sum of all items gives the total score which ranges from 0 to 48. The cut off score of 19 is suggestive for a clinically relevant case of perceived injustice.
  This questionnaire obtains two correlated factors: severity/irreparability of loss and blame/unfairness. The Dutch version of the IEQ has good (test-retest) reliability (ICC = 0.86-0.87). The scores obtained using the IEQ are valid.
Health care utilization (HCU) | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Medical consumption, the type, dose, method of administration and frequency of analgesic, NSAID or symptom-modifying medication, as well as surgeries will be recorded. Health care use will be evaluated using the combination of three questionnaires (online):
  1. the Medical Consumption Questionnaire (MCQ)
  2. the Productivity Cost Questionnaire (PCQ)
  3. the EuroQol EQ-5D
  The combination of these questionnaires is advised by the Institute for Medical Technology Assessment, Erasmus University Rotterdam (the Netherlands).

OTHER OUTCOMES:
Sleep quality | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Pittsburgh Sleep Quality Index (PSQI): is a self-rated questionnaire to measure sleep quality and disturbance over 1 month. It is based on 19 items which generate a global score, ranging between 0 and 21, and 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores above 5 signifies a poor sleeper. It is a reliable and valid measurement tool and internal consistency is acceptable in breast cancer population (Cronbach's alpha = 0.80).
Sleep insomnia | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Insomnia Severity Index (ISI): is a questionnaire to detect cases of insomnia and asses the insomnia severity of both night-time and daytime components of insomnia. It is based on 7 items measured on a 5-point Likert scale (0-4) which generates a total score ranging from 0 (no insomnia) to 28 (great insomnia severity). The cut-off score of 10 is optimal for detecting insomnia cases and a change score of -8.4 points is associated with a moderate improvement. ISI is a valid and reliable instrument in cancer patients and had an adequate concurrent validity of (r = 0,65).
Fatigue severity | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Fatigue Severity Scale (FSS): is used to evaluate global fatigue severity in a number of chronic medical conditions such as palliative cancer. It is a short questionnaire with 9-items and the total score ranges between 9 (no fatigue) and 63 (maximum fatigue). The FSS is a reliable and valid measurement in cancer patients. The internal consistency of the FSS is highly acceptable (Cronbach's alpha = 0.96).
Pain catastrophizing | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Pain Catastrophizing Scale (PCS): is a self-reported questionnaire to assess catastrophic thoughts or feelings accompanying the previously experienced pain. It is a 13-item measure that evaluates 3 subscales of catastrophizing: rumination, magnification and helplessness on a 5-point Likert scale. This scale ranges from 0 (not at all) to 4 (all the time) with a total score between 0 and 52. The PCS factor scales are valid and reliable.
Pain cognitions | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Brief Illness Perceptions Questionnaire-Dutch Language Version (Brief IPQ-DLV): measures five illness perceptions and consists nine items. Five items assess cognitive illness (consequences, personal control, treatment control and identity), two items assess emotional perceptions (concern and emotions), one item assesses illness comprehensibility and one item assesses causal perception. The first eight items are rated on a 10-point Likert scale and the ninth item is rated as an open-ended question which asks to list three most important causal factors in the illness. The Brief IPQ-DLV has acceptable psychometric properties. The Smallest Detectable Change (SDC) is 3 point for item 1 to 8.
Pain behaviour | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Pain Vigilance and Awareness Questionnaire (PVAQ): is designed to consider behaviour over the last 2 weeks in chronic pain patients. It consists 16-items that assesses attention to pain. The frequency of each item is rated on a 6-point Likert scale ranging from 0 (never) to 5 (always) with a total score ranges between 0 and 90. The higher the score, the more suggestive for a higher degree of vigilance and awareness to pain. It is highly correlated with pain-related measures such as catastrophizing, and weakly correlated with measures of unrelated constructs, such as trait anxiety. The PVAQ is a reliable and valid measurement in chronic patients.
Depression, Anxiety, Stress | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Depression, Anxiety, Stress Scale 21 items (DASS-21): is an instrument that is used to assess anxiety and depression. Twenty-one items are subdivided in 3 categories: depression (7 items), anxiety (7 items) and stress (7 items). Each item is scored on a 4-point Likert scale ranging from 0 (not at all) to 3 (most of the time). The higher the item score, the more severe symptom of psychological distress is identified. The total score, used for the interpretation, is the sum of all items multiplied by two. The DASS-21 is a valid and reliable assessment tool in cancer patients.
Anger | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  State-Trait Anger Expression Inventory-II (STAXI-II): is a self-reported 57-item questionnaire that assesses the level and frequency of anger experience, expression and control. It consists three parts: (a) how angry the examinee currently feels, (b) how angry the examinee generally feels, and (c) how the examinee reacts when angry. Every item in each subscale is assessed on a 4-point Likert-scale. The validity and reliability of the STAXI-II questionnaire are satisfactory supported.
Acceptance | T0: within the week before the randomisation and the start of the intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Acceptance and Action Questionnaire - II (AAQ-II): is a self-reported 7-item questionnaire that assesses the amount of acceptance and experiential avoidance, or its opposite: psychological flexibility. Every item is a statement that is scored on a 7-point Likert-scale in which one can indicate to what extent these are applicable. The higher the total score, the lower the acceptance and the higher the experiential avoidance. The psychometric qualities of the Dutch translation of the AAQ-II are good with an internal reliability of 0.87 and a construct validity of -0.67 to -0.79 for oppression and psychological complaints.
Treatment adherence and compliance | During intervention period (after T0 and before T1)
  Patients' attendance at treatment sessions will be recorded. Patient adherence for the treatment sessions will be calculated as the ratio of the number of treatment sessions that were actually carried out versus the number of prescribed sessions. For the home sessions (incl. working with the information leaflet), patients will be asked to record the sessions' content in a personal log book. Treatment adherence will be calculated as a ratio of the number of sessions that were actually carried out at home versus the total number of prescribed home sessions. Patient drop-out and the reason for withdrawal will be registered.
Co-interventions | T0: within the week before randomisation and start of intervention; during intervention; T1: immediately after completing intervention; T2: 6 months after therapy completion; T3: 12 months after therapy completion; T4: 24 months after therapy completion
  Co-interventions will be closely monitored. Medical consumption, including the type, dose, method of administration and frequency of medication, as well as any other interventions will be recorded.
Personal characteristics | T0: within the week before the randomisation and the start of the intervention
  Personal characteristics including date of birth, nationality, race/ethnicity, level of education, professional situation, family income, relationship status, physical activity, smoking status, alcohol consumption, Body Mass Index (BMI), comorbidities, lymphedema, type of surgery, hormone therapy, chemotherapy, radiotherapy, immunotherapy, time since onset of complaints, time since complement of treatment, and treatment expectations will be collected at baseline.
Screening dementia or cognitive impairment | During screening period; before T0
  Participants will be excluded if they are suffering from dementia or cognitive impairment (unable to understand the test instructions and/or a result of ≤11, corresponding with MMSE ≤23, on the Six-item Cognitive Impairment Test (6-item CIT) is a short questionnaire containing 6 items.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (4):
- Belgium (4):
  - AZ Rivierenland, Bornem, Antwerpen
  - Vrije Universiteit Brussel, Jette, Brussels Capital
  - Universiteit Hasselt - campus Diepenbeek, Diepenbeek, Limburg
  - Imeldaziekenhuis, Bonheiden, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: Yes
After the project, the data will be archived in the VUB University Archive with restricted access. Data sharing is only permitted if all involved parties agree, and a Data Sharing Agreement has been signed.
  Open Access will not be possible due to the high degree of confidentiality of the pseudonymized medical data, although all requests regarding sharing the research data will be considered by the parties.
  The university server is equipped with user-level access permission management. Participants' personal data will be coded, and system encryption will be used to protect the coded data.
  No costs are expected, but project and/or research group funds will cover any potential data sharing costs.
Supporting Information: Study Protocol
Time Frame: The generated research data (both raw and processed data), the accompanying metadata and all documentation necessary to reuse the data will be transferred to the VUB University Archive server (K-drive) designed for long-term data archiving (managed by VUB ICTS with automatic back-up procedures).
  We will adhere to the principle of preservation of data and the policy of VUB (Vrije Universiteit Brussel) is to use a preservation term of 10 years, which we will apply.
  Data will be available upon publication of the research results until 10 years after.
Access Criteria: Upon request by mail

REFERENCES:
- [Derived] Roose E, Van Bogaert W, Mostaqim K, Huysmans E, Nijs J, van Wilgen CP, Beckwee D, Timmermans A, Fontaine C, Lahousse A. An exploration of the relationship between perceived injustice and pain severity in breast cancer survivors: a structural equation model. Support Care Cancer. 2025 Jul 9;33(8):670. doi: 10.1007/s00520-025-09655-8. PMID 40629158
- [Derived] Roose E, Huysmans E, Leysen L, Mostaqim K, Van Wilgen P, Beckwee D, De Couck M, Timmermans A, Bults R, Nijs J, Lahousse A. Effect of perceived injustice-targeted pain neuroscience education compared with biomedically focused education in breast cancer survivors: a study protocol for a multicentre randomised controlled trial (BCS-PI trial). BMJ Open. 2024 Jan 17;14(1):e075779. doi: 10.1136/bmjopen-2023-075779. PMID 38233049